CLINICAL TRIAL: NCT04418882
Title: Septic Management and Outcome of Open Fracture : a 7 Years Retrospective Cohort Study
Brief Title: Septic Management and Outcome of Open Fracture
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20-204
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Open Fracture; Pseudarthrosis; Bone and Joint Infection
Keywords: bone and joint infection; Pseudarthrosis; Open Fracture
MeSH Terms: conditions — Fractures, Open; Pseudarthrosis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non septic open fracture: patients having had an open fracture without septic evolution
  Interventions: Other: management and follow up of all open fractures
- septic open fracture: patients having had an open fracture with septic evolution
  Interventions: Other: management and follow up of all open fractures

INTERVENTIONS:
Other: management and follow up of all open fractures — to evaluate the development of sepsis after an open fracture and then, if there is a development of a pseudarthrosis too.

SUMMARY:
The aim is the study of the management and outcome of the open fractures.

Some open fractures will become pseudarthrosis. Thoses pseudarthrosis may be septic or not.

The management and evolution of all the open fractures will be described in order to identify the presence or not of a sepsis and then a development of a pseudarthrosis (septic or non septic).

ELIGIBILITY:
Inclusion Criteria:

* all patients with open fractures

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had an open fractures managed at the HCL
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
description of non septic open fracture | 24 months
  description of surgical management
description of patients with non septic open fracture | 1 month
  description of patients : average age, medical background
description of septic open fracture : bacteriology | 24 months
  type of bacteria involved in the infection
description of septic open fracture : evolution | 24 months
  description of symptoms
description of septic open fracture : management | 24 months
  description of surgical and medical management
description of septic open fracture : patients | 24 months
  description of patients : average age, medical background
description of pseudarthrosis: symptoms | 24 months
  description of symptoms
description of pseudarthrosis : management | 24 months
  description of management: surgical and medical management
description of septic pseudarthrosis : patients | 24 months
  description of patients : average age, medical background
description of septic pseudarthrosis : bacteriology | 24 months
  type of bacteria involved in the infection
treatment failure | 24 months
  rate and description of treatment failure.Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr